CLINICAL TRIAL: NCT03451240
Title: A Mixed Methods Evaluation of HPI Resilience Intervention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Health and Wellness Solutions, Inc. (Industry)
Collaborators: Lake Nona Institute (Unknown); Grounded Solutions Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017-07A
Record Dates: First submitted 2018-02-05; First posted 2018-03-01 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Stress
Keywords: Stress; Resilience

STUDY DESIGN:
Intervention Model Description: To determine the impact of the Corporate Athlete® Resilience product through recalibrating mindset and changing resilience supportive behavior.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Behavioral: Corporate Athlete® Resilience

INTERVENTIONS:
Behavioral: Corporate Athlete® Resilience — The product Corporate Athlete® Resilience Training Program ("CAR Training"), is a one day training program aimed to educate participants about stress management and stress recovery techniques.
  The content of the training program is divided into two parts:
  1. Introduction to stress and resilience: an overview of stress and its impact on wellbeing, combined with the definition of resilience and its linking to daily performance.
  2. Introduction and implementation of stress management and resilience techniques: an overview of applicable stress management and resilience tools, combined with real time application methods. These activities aim to help individuals recover and grow from a stressful state into meaningful life engagement. The desired overall effect is better performance at home and at work.

SUMMARY:
The primary objective of the Resilience Study is to determine the impact of the Corporate Athlete® Resilience product through recalibrating mindset and changing resilience supportive behavior.

Analysis will be performed via Survey and Study Interviews (two methods) to determine how the CAR Training recalibrated and impacted the Research Participants mindset and resilience state.

1. Tool: Stress Mindset Measure-General (SMM-G)

Additional analysis will evaluate participants' engagement in behavior changes in the first 30 days.

2. Tool: Energy Management Behaviors.

Secondary objectives include further analysis to determine if the intervention group demonstrated significant improvements in the following measures:

1. Brief Resilience Scale (BRS)

2. Public Health Surveillance Wellbeing (PHS-WB)

3. Sleep Habits (Rand MOS)

4. Health, Wellbeing and Productivity (SF36, HPQ)

5. Work Productivity and Activity Impairment (WPAI)

6. Brief Cope

7. Perceived Stress (PSS)

In addition, demographic assessments will be collected.

DETAILED DESCRIPTION:
Methodology: This is an interventional mixed methods (qualitative & quantitative) study, with pre-post design for research participants in one session. All participants will be measured at two time points: surveys will be collected between 3-weeks to the day of intervention for baseline, 1-month post intervention.

In addition, Qualitative interviews will be conducted on a rolling basis between 3-60 days post intervention. The qualitative portion is a semi-structured interview will be conducted with the purpose of understanding how participants recalibrated their mindset and impacting their resilience behaviors.

Study Advertisement combined with the Resilience Program Advertisement will be posted by the Lake Nona Institute. Potential Research Participants will be self-selected, and will contact the Lake Nona Study Coordinator for additional information. The self-selected individuals will receive HPI materials via mail, in addition to Study and Resilience Program eligibility information.

Potential Research Participants will undergo Screening and Consenting procedures at the Lake Nona Institute. The Research Participant will be required to sign and date a paper based Informed Consent Document, and provide additional contact information, such as individual email address, phone number etc.

Enrolled Research Participants will be scheduled to attend the CAR Training Session.

On the day of the CAR Training, the Research Participants will receive a set of questionnaires as part of the Corporate Athlete® Resilience Program ("HPI Questionnaire"), in addition to a set of Study Specific Questionnaires ("Study Questionnaire"). A description study activities ("Study Guide") and a description of session activities ("Agenda") consists of the introduction to stress and resilience session, will be distributed to all Research Participants.

30 days following the CAR Training, the Research Participants will receive a follow-up HPI questionnaires and a Study questionnaires which will be utilized in the Resilience Research Study Analysis.

3-60 days upon completion of the CAR Training, the Research Participants will be asked to complete a Research Study Qualitative Telephone, Video or Face-to-Face Interview ("Study Interview").

ELIGIBILITY:
Inclusion Criteria:

1. Be an adult (18 years or older);
2. Be a participant in the LNLP (i.e., provided consent for the project);
3. Meet =>2 stress experience level parameters on Stress Mindset Measure-General (SMM-G);
4. Meet =< 4.3 on the Brief Resilience Scale (BRS);
5. Be willing to attend a full day training program at the Lake Nona Institute during the designated training date;
6. Be willing to provide email and phone number as a contact method;
7. Must speak, read, and understand English fluently;
8. Be able to comprehend and follow the requirements of the study;
9. Research Participant must have a valid e-mail address;
10. Be able to provide Informed Consent;
11. Be willing and able to comply with all study procedures for the duration of the study.

Exclusion Criteria:

1. Is not an adult (18 years or older);
2. Has not consented to participate in the LNLP;
3. Does not meet the stress or resilience parameters (as defined above);
4. Unwilling or unable to provide consent and sign the ICF;
5. Unwilling or unable to complete study related questionnaires;
6. Have a physical or cognitive impairment that would interfere with their ability to provide accurate information;
7. Not able to speak, read, or understand English fluently.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-09-16 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Stress Mindset Measure-General (SMM-G) | 3-weeks to the day of intervention for baseline, 1-month post intervention (assessing for a change)
  The Stress Mindset Measure-General (SMM-G) is an 8-item measure developed to address the extent to which an individual adopts a mindset that the effects of stress are enhancing or debilitating.
Energy Management Behaviors | 3-weeks to the day of intervention for baseline, 1-month post intervention (assessing for a change)
  The Energy Management Behaviors (EMB) assessment tool consists of 40 items measuring the impact of an individual's behavior, their desired life changes as well as their stress, recovery and energy.
Qualitative Interviews | 3-60 days post intervention
  A qualitative telephone or video interview where the grounded theory research method will be used to understand 'the phenomena that occur across participants'. The purpose is to understand how participants recalibrate their mindsets and the impact of recalibration on their resilience behaviours following attendance at a one day training event.

SECONDARY OUTCOMES:
Brief Resilience Scale (BRS) | 3-weeks to the day of intervention for baseline, 1-month post intervention
  The Brief Resilience Scale (BRS) is a 6-item measure created to assess the ability to bounce back or recover from stress. It is scored by reverse coding items 2, 4, and 6 and finding the mean of the six items. A higher score equals higher resilience.
Public Health Surveillance Wellbeing (PHS-WB) | 3-weeks to the day of intervention for baseline, 1-month post intervention
  The Public Health Surveillance Well-Being Scale (PHS-WB) comprises 10-items guaging self-reported mental, physical, and social components of well-being. Response options for 6 of the items are on a 5-point Likert-type scale. The responses options range from "strongly disagree" to "strongly agree," "none of the time" to "all of the time," and "poor" to "excellent." Three of the items are based on a 10-point Likert-type scale. Response options for the 10-point items range from "very dissatisfied" to "very satisfied." One item assesses energy/vitality over the past 30 day. The responses for that item ranged from 0 to 30. A score for the PHS-WB scale was created by summing the 10 items for each respondent.
Sleep Habits (Rand MOS) | 3-weeks to the day of intervention for baseline, 1-month post intervention
  The MOS Sleep Scale is a 12-item instrument, which measures multiple facets of sleep. The MOS Sleep Scale yields a sleep problems index and six scale scores: sleep disturbance (have trouble falling asleep, how long to fall asleep, sleep was not quiet, awaken during your sleep time, and have trouble falling asleep again), sleep adequacy (get enough sleep to feel rested upon waking in the morning and get amount of sleep needed), daytime somnolence (drowsy during day, have trouble staying awake during the day, and take naps), snoring, awaken short of breath or with headache, and quantity of sleep. Quantity of sleep is scored as the average hours slept per night. The other scales and problems index are scored on a range from 0 to 100 with higher scores indicating more of the concept being measured.
Health, Wellbeing and Productivity (SF36, HPQ) | 3-weeks to the day of intervention for baseline, 1-month post intervention
  The SF-36 is a 36-item questionnaire which measures QoL across eight domains, which are both physically- and emotionally-based. The eight domains that the SF-36 measures are as follows: physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, and general health.
Work Productivity and Activity Impairment (WPAI) | between 3-weeks to the day of intervention for baseline, 1-month post intervention
  The WPAI:GH is a six-item questionnaire, measuring the effect of one's health problems on their ability to work and perform regular activities. The questions have four scores: (1) percentage work time missed due to health (absenteeism); (2) percentage impairment at work due to health (presenteeism); (3) percentage overall work productivity loss due to health (absenteeism and presenteeism); and (4) percentage daily activity impairment outside of work due to health. Higher scores indicate prolonged sick leave or impairment and decreased productivity.
Brief Cope | 3-weeks to the day of intervention for baseline, 1-month post intervention
  The Brief COPE inventory is a 28-item measure used to assess ways that an individual copes with stress in their life, in particular around the time a stressful event has occurred.
Perceived Stress (PSS) | 3-weeks to the day of intervention for baseline, 1-month post intervention
  The Perceived Stress Scale (PSS) is a 10-item scale used to measure the perception of stress, specifically, the degree which situations in one's life are appraised as stressful.The total score is calculated by finding the sum of 10 items, reverse coding questions 4, 5, 7, & 8. The PSS has a range of scores between 0 (no stress) and 40 (high stress). A higher score indicates more stress.

CONTACTS AND LOCATIONS:
Overall Officials: Shawn Mason, PhD, Principal Investigator — Johnson & Johnson Health and Wellness Solutions
Locations (1):
- The Human Performance Institute, Orlando, Florida, United States